CLINICAL TRIAL: NCT06764134
Title: Study Protocol for an Investigator Initiated, Observational Prospective Study, Evaluating the Rate of Postoperative Pancreatic Fistula in Distal Pancreatectomy Using AEON™ Endostapler
Brief Title: Assessing Pancreatic Fistula Rates After Distal Pancreatectomy Using AEON Endostapler
Acronym: AEON-DP
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Arianeb Mehrabi, MD, Professor, University Hospital Heidelberg
Other Study IDs: S-473/2024
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pancreas; Fistula; Pancreas Cancer; Pancreatic Disease; Surgery-Complications; Surgery
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective, observational study evaluates the rate of postoperative pancreatic fistula (POPF) following distal pancreatectomy (DP) using the AEON™ Endostapler. The study involves 110 patients undergoing DP and assesses primary outcomes based on the International Study Group of Pancreatic Fistula (ISGPF) classification, alongside secondary perioperative parameters. The findings aim to optimize surgical techniques, reduce complications, and improve healthcare outcomes.

DETAILED DESCRIPTION:
This is a prospective, observational, monocentric study designed to evaluate the incidence of postoperative pancreatic fistula (POPF) following distal pancreatectomy (DP) performed using the AEON™ Endostapler. POPF is one of the most serious complications after DP, and effective stump closure remains a critical challenge in reducing its occurrence. The study will involve 110 patients who meet the inclusion criteria and undergo DP at the University of Heidelberg.

Primary outcomes will focus on the rate of clinically relevant POPF as defined by the International Study Group of Pancreatic Fistula (ISGPF). Secondary outcomes include intraoperative and postoperative parameters, such as estimated blood loss, operation duration, ICU and hospital stay, reoperation rates, and 90-day mortality. All outcomes will be assessed following standardized protocols.

Patients will be enrolled after providing informed consent and will receive follow-up evaluations at specific time points, including postoperative days 1, 3, 14, 30, and 90. Amylase levels in drain fluid will be measured to monitor pancreatic leakage. Data collected during the study will be analyzed to assess the effectiveness and safety of the AEON™ Endostapler in reducing POPF and other complications.

The findings aim to contribute critical evidence to improve surgical practices and outcomes for DP patients, potentially shaping future guidelines and reducing healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Ability to understand the nature and consequences of the study.
* Provision of written informed consent.
* Scheduled for minimally invasive or open distal pancreatectomy (DP) for any indication, with or without splenectomy and/or left adrenalectomy.

Exclusion Criteria:

* Inability to comply with study procedures or follow-up.
* Multivisceral resection beyond left adrenalectomy.
* History of previous pancreatic surgeries.
* Expected lack of compliance with the study protocol.
* Participation in another trial that may interfere with the intervention or outcomes of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 years or older scheduled to undergo minimally invasive or open distal pancreatectomy (DP) for any indication, with or without splenectomy and/or left adrenalectomy. These patients will be recruited from the University of Heidelberg and screened for eligibility based on inclusion and exclusion criteria. Participants must provide informed consent and demonstrate the ability to comply with study procedures and follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Clinically Relevant Postoperative Pancreatic Fistula (POPF) | Up to 90 days post-surgery.
  The rate of clinically relevant POPF will be assessed based on the International Study Group of Pancreatic Fistula (ISGPF) definition, which includes drain output of any measurable volume of fluid on or after postoperative day 3 with an amylase content exceeding three times the upper limit of normal serum amylase activity, associated with a clinically relevant condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Baden-Wurttemberg, Germany